CLINICAL TRIAL: NCT03962153
Title: New Ultrasonographic Parameters for Fetal Weight Prediction
Brief Title: Ultrasonographic Parameters for Fetal Weight Prediction
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Pasquale De Franciscis, Associate Professor, University of Campania Luigi Vanvitelli
Other Study IDs: N.603
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Fetal Growth Abnormality
Keywords: fetal growth; ultrasonographic parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Obstetric Ultrasonography — Obstetric Ultrasonography

SUMMARY:
The hypothesis is to increase the predictability of the ultrasound examination evaluating new fetal parameters: in fact the thickness of the soft tissues can contribute significantly to the fetal weight and the characteristics of the thoracic cage may correlate with the fetal weight.

DETAILED DESCRIPTION:
Estimation of fetal weight (EFW: Estimated Fetal Weight) with ultrasound examination is a common practice in obstetrics and is important for planning the mode and timing of birth, especially in pregnancies at risk for altered fetal growth.

The conditions most commonly associated with impaired fetal growth are:

* IUGR: in these cases the ultrasound estimate of fetal weight is fundamental to decide the timing of delivery, since the neonatal outcome correlates positively with the fetal weight as well as with the flowmetry parameters
* fetal macrosomia (fetal weight greater than 4500 g) associated or not with gestational diabetes: in such cases an accurate estimation of the fetal weight is necessary and careful evaluation of any fetal-pelvic disproportion to decide both the timing of the birth that can be anticipated compared to at the physiological end of pregnancy is the mode of birth, vaginal or laparotomic in the event of a pelvic fetus disproportion.

In the 1970s the estimate of fetal weight was based on the measurement of the symphysis-fundus uterine distance (SFH) for which:

* SFH <33 cm: predictive of a fetal weight <3100 gr
* SFH> 34 cm: predictive of a fetal weight = o> 4000 gr.

At present, the fetal weight estimate is performed with biometric ultrasound parameters:

* DBP: biparietal diameter
* HC: head circumference
* AC: abdominal circumference
* FL: femur length There are standardized tables of variation of these parameters according to the gestational epoch for which the knowledge of the correct gestational epoch is fundamental for the correct interpretation of the data.

The fetal weight is calculated using mathematical formulas automatically obtained from ultrasound equipment of which the most used:

* Shepard's formula as a function of BPD and AC.
* formula of Campbell and Wilkin: it is in function of the abdominal circumference
* Hadlock formula: use the combination of different biometric parameters (BPD-HC-AC-FL).

Even if the guidelines provide for three ultrasound examinations for physiological pregnancies (one for each trimester of pregnancy), it is common practice to evaluate the biometric ultrasound parameters at the end of pregnancy and in any case when the patient is admitted for the delivery. It is obvious that in this time of pregnancy a closer correlation between biometric parameters and fetal weight is observed.

The problems related to the ultrasound estimation of fetal weight are represented by:

* significant intra-operator variability
* reduced accuracy for extremes of fetal weight (small or macrosomic fetuses)
* about 10% discrepancy between estimated fetal weight on an echographic basis according to Hadlock and actual weight of the newborn at birth.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* fetal structural and / or chromosomal anomalies
* multiple pregnancies
* premature births (gestational age <37w)

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: single pregnancies, free of complications, with delivery completed between 37 and 42 weeks, but within a week of the last ultrasound examination performed. Patients are selected among those candidates with elective caesarean section, pregnant who come to hospital for prodroma of labor and conditions that require induction of childbirth such as prolonged pregnancy or PROM.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
biparietal diameter | 9 months
  Evaluation of biparietal diameter
head circumference | 9 months
  evaluation of head circumference
abdominal circumference | 9 months
  Evaluation of abdominal circumference
femur length | 9 months
  Evaluation of femur length
transtentorial diameter | 9 months
  Evaluation of transtentorial diameter
distance between L1-L4 lumbar vertebrae | 9 months
  Evaluation of distance between L1-L4
Fetal Weight | 9 months
  Evaluation of Fetal Weight

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Woman, Child and General and Specialized Surgery, University of Campania "Luigi Vanvitelli", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No